CLINICAL TRIAL: NCT06999200
Title: Evaluation of the Effectiveness of Subcutaneous and Intracutaneous Local Anesthesia for Postoperative Analgesia in Patients Undergoing Cesarean Section Under General Anesthesia: a Prospective Randomized Controlled Trial (RCT)
Brief Title: Neural Therapy in Cesareans
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Yilmaz Guler, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: NT-2016
Record Dates: First submitted 2025-05-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Visual Analogue Scale
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subcutaneous local anesthesia group: who received subcutaneous local anesthesia at the end of C/S surgery
  Interventions: Drug: neural therapy
- Intracutaneous local anesthesia group: who received intracutaneous local anesthesia at the end of C/S surgery
  Interventions: Drug: neural therapy
- Parenteral analgesia group: who received parenteral analgesia after C/S surgery
  Interventions: Drug: neural therapy

INTERVENTIONS:
Drug: neural therapy — This prospective study will be conducted with mothers who underwent general anesthesia for labor or elective cesarean delivery and local anesthesia for postoperative pain management during a one-year period following ethical approval.

SUMMARY:
In the management of pain after Caesarean section (C/S), opioid or nonsteroidal anti-inflammatory parenteral drugs are applied. These drugs are insufficient in some cases and may cause pain attacks during the day. Higher doses and repeated drug applications or combined drug administration may cause drug side effects and interactions. Alternative applications to provide analgesia include subcutaneous and intracutaneous local anesthetic application to the wound site. Although the effectiveness of these applications has been tested in individuals with different clinical characteristics and has been shown to be largely more successful, they have not been sufficiently introduced into routine practice. There is a need to review the pain methods suggested in the literature and develop new solutions that can be applied more optimally, improve the patient's pain management in the postoperative period, and increase their quality of life and satisfaction.

It aims to evaluate the success of subcutaneous and intracutaneous local anesthesia applications compared to traditional applications, and to find the most optimal management.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy,
* Term (>37 weeks) and preterm (28-34 weeks) pregnancy,
* Cases that received general anesthesia for cesarean section,
* Cases with and without labor,
* Cases with and without obesity,
* Cases that had their first or second cesarean section

Exclusion Criteria:

* Pregnant women under 19 years of age,
* Those with a history of allergic reactions to analgesics to be used,
* Stillbirth,
* Surgical complications during C/S and placement of an abdominal drain,
* No head or breech presentation during C/S,
* Occiput posterior presentation during C/S,
* Anhydramnios and polyhydramnios,
* Allergic reactions to the drugs used in the study, alcohol dependence, drug and substance dependence, chronic pain syndrome, neuropathic pain disorder history,
* History of clinically significant cardiovascular, pulmonary, hepatic, renal, neurological, psychiatric, metabolic disease.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women aged 19-45 who underwent a caesarean section under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 48 hours
  1=no pain, 10=worst pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reed SE, Tan HS, Fuller ME, Krishnamoorthy V, Ohnuma T, Raghunathan K, Habib AS. Analgesia After Cesarean Delivery in the United States 2008-2018: A Retrospective Cohort Study. Anesth Analg. 2021 Dec 1;133(6):1550-1558. doi: 10.1213/ANE.0000000000005587. PMID 34014182
- [Result] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462